CLINICAL TRIAL: NCT02297906
Title: Pharmacokinetics of Intranasal Ketorolac in Children
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrolment issues
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Assistant Professor of Pediatrics at CUMC, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAN5404
Record Dates: First submitted 2014-11-14; First posted 2014-11-21 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Evaluating Pharmacokinetics of Intranasal Ketorolac; Pain
Keywords: Intranasal; Ketorolac; Pharmacokinetics; Pediatric
MeSH Terms: conditions — Pain | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal ketorolac (Experimental): Ketorolac 0.5 mg/kg, maximum single dose = 30 mg. Administered once by intranasal route using a mucosal atomization device.
  Interventions: Drug: Ketorolac
- Intravenous ketorolac (Active Comparator): Ketorolac 0.5 mg/kg, maximum single dose = 30 mg. Administered once by intravenous route.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — Non-steroidal anti-inflammatory drug
  Other Names: Toradol

SUMMARY:
Ketorolac is a non-steroidal anti-inflammatory drug (NSAID) that is typically given to both adults and children by the intravenous (IV) or intramuscular (IM) route for analgesic purposes. Ketorolac can also be given by the intranasal (IN) route using a mucosal atomization device (MAD). We aim to study the pharmacokinetics of ketorolac when administered by the IN route using the MAD.

DETAILED DESCRIPTION:
The intranasal (IN) route of administering medications is an effective means of delivering analgesics to children in a painless and minimally distressing manner, especially in comparison to traditional means of intravenous (IV) or intramuscular (IM) administration, which require a painful and distressing needle stick.

Ketorolac is an analgesic that is commonly administered to children, and can be given by the IN route, in addition to the IV and IM routes. However, the pharmacokinetics of intranasal ketorolac when administered in children has only been described in a limited fashion. The administration of IN ketorolac in children, using the proprietary SPRIX device, which atomizes a fixed amount of ketorolac, produces serum concentrations of ketorolac that are associated with analgesia. However, the concentrations of ketorolac achieved using a mucosal atomization device (MAD) has not yet been evaluated in children presenting to the emergency department. The MAD is a plastic device that attaches to the top of a syringe (see figure). The MAD is much more commonly used for atomizing medications; allows a variable dosage to be administered; and has been shown to be a means of effectively delivering other analgesics and sedatives intranasally.

The purpose of this study is to assess the pharmacokinetics of IN ketorolac when using a MAD to deliver the medication in children presenting to the emergency department. We will determine the maximum serum concentration achieved (Cmax), time to maximum serum concentration achieved (Tmax), and bioavailability (compared to IV ketorolac) when ketorolac is administered intranasally using a MAD.

ELIGIBILITY:
Inclusion Criteria:

* Present to the emergency department with a painful condition for which the treating physician decides to administer ketorolac as part of their usual care.

Exclusion Criteria:

* Known allergy to ketorolac
* Contraindication to receiving ketorolac
* Receiving any NSAID within the past 6 hours
* Presence of an intranasal obstruction that cannot be readily cleared using suction or nose-blowing
* Inability to speak English or Spanish
* Critical illness

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Cmax of intranasal ketorolac | 60 minutes
  Maximum serum concentration of ketorolac, after intranasal administration

SECONDARY OUTCOMES:
Tmax of intranasal ketorolac | 6 hours
  Time to maximum serum concentration of ketorolac, after intranasal administration
Bioavailability of intranasal ketorolac | 6 hours
  Bioavailability of intranasal ketorolac; expressed as a percentage (numerator = serum levels achieved by intranasal administration, denominator = serum levels achieved by intravenous administration)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Tsze, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian Morgan Stanley Children's Hospital, New York, New York, United States